CLINICAL TRIAL: NCT03671265
Title: A Single Arm Exploratory Study of Chemotherapy Plus Radiation Therapy and Anti-PD-1 Antibody SHR-1210 in Treating Patients With Locally Advanced Esophageal Squamous Cell Carcinomas
Brief Title: Combination of Chemotherapy Plus RT and SHR-1210 to Treat Patients With ESCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-CRT-ESC-IIT
Record Dates: First submitted 2018-09-02; First posted 2018-09-14 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2018-08

CONDITIONS: Esophageal Cancer
Keywords: Esophageal Cancer; Concurrent chemoradiation; Immunotherapy; SHR-1210; Apatinib
MeSH Terms: conditions — Esophageal Neoplasms | interventions — camrelizumab; spartalizumab; Radiotherapy, Intensity-Modulated; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1210 + Chemotherapy + Radiotherapy (Experimental): Radiotherapy(IMRT or VMAT): 95%PTV 54Gy/30 fraction,95%PTV 60Gy/30 fraction ,5 fractions per week, for 6 weeks. Radiation begun the day on which first dose of SHR-1210.
  SHR-1210 (200mg fixed dose every 2 weeks, one cycle is four weeks, total 8 cycles ) will be administered as an intravenous infusion over 30 minutes.
  Chemotherapy: Docetaxel 25mg/m2/w, intravenous infusion on days 1, 8, 15, 22, total 4 cycles; Cisplatin 25mg/m2/w, intravenous infusion on days 1, 8, 15, 22;, total 4 cycles.
  Apatinib: 250mg/d，PO Qd(4 weeks after Radiotherapy, until the end of 8th ycle )
  Interventions: Drug: SHR-1210; Radiation: IMRT or VMAT; Drug: Apatinib

INTERVENTIONS:
Drug: SHR-1210 — SHR-1210 is a humanized anti-PD1 IgG4 monoclonal antibody.
  Other Names: Anti-PD-1 Antibody
Radiation: IMRT or VMAT — The IMRT or VMAT technique was used in our study.
Drug: Apatinib — Apatinib is a small molecule tyrosine kinase inhibitor targeting vascular endothelial growth factor receptor-2.

SUMMARY:
SHR-1210 is a humanized anti-PD1 IgG4 monoclonal antibody. This is an openlabel，single center ，non-randomized ，Single Arm Exploratory Study . This clinical study is an investigator-initiated clinical trial（IIT). The objective of this study is to evaluate the efficacy and safety of radiation therapy combined with anti-PD-1 antibody SHR-1210 and chemotherapy in patients with Locally Advanced Esophageal Squamous Cell Carcinomas。

ELIGIBILITY:
Inclusion Criteria:

1. age:18-75 years, male or female.
2. Histologically confirmed primary Squamous Cell Carcinoma of the Esophagus,Local advanced esophageal cancer diagnosed by pathology and imaging,clinical stage T3-4N0M0, T1-4N+M0,Ⅱ-Ⅳa.
3. Pre-treatment evaluation can not tolerate concurrent radiochemotherapy or rejection of the concurrent use of chemotherapy with radiotherapy.
4. Measurable disease based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
5. ECOG 0-1.
6. Adequate organ function.
7. Life expectancy of greater than 6 months.
8. Patient has given written informed consent.

Exclusion Criteria:

1. Patients who have or are currently undergoing additional chemotherapy, radiation therapy, targeted therapy or immunotherapy.
2. Known history of hypersensitivity to macromolecular protein preparation or any components of the SHR- 1210 formulation.
3. Subjects before or at the same time with other malignant tumors (except which has cured skin basal cell carcinoma and cervical carcinoma in situ);
4. Subjects with any active autoimmune disease or history of autoimmune disease

   - Page 4 of 4 [DRAFT] -
5. Uncontrolled clinically significant heart disease, including but not limited to the following: (1) > NYHA II congestive heart failure; (2) unstable angina, (3) myocardial infarction within the past 1 year; (4) clinically significant supraventricular arrhythmia or ventricular arrhythmia requirement for treatment or intervention;
6. Active infection or an unexplained fever > 38.5°C during screening or before the first scheduled day of dosing (subjects with tumor fever may be enrolled at the discretion of the investigator);
7. Received a live vaccine within 4 weeks of the first dose of study medication.
8. Pregnancy or breast feeding.
9. Decision of unsuitableness by principal investigator or physician-incharge.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AE), Serious Adverse Event(SAE) Adverse events | Through study completion, an average of half a year]
  Incidence of Treatment-Emergent Adverse Events

SECONDARY OUTCOMES:
ORR | Through study completion, an average of 1 year
  Objective Response Rate
PFS | 1year and 3years
  Progression-Free Survival
OS | 1year and 3years
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Yan C, Huang H, Zheng Z, Ma X, Zhao G, Zhang T, Chen X, Cao F, Wei H, Dong J, Tang P, Jiang H, Wang M, Wang P, Pang Q, Zhang W. Spatial distribution of tumor-infiltrating T cells indicated immune response status under chemoradiotherapy plus PD-1 blockade in esophageal cancer. Front Immunol. 2023 May 19;14:1138054. doi: 10.3389/fimmu.2023.1138054. eCollection 2023. PMID 37275884
- [Derived] Ma X, Guo Z, Wei X, Zhao G, Han D, Zhang T, Chen X, Cao F, Dong J, Zhao L, Yuan Z, Wang P, Pang Q, Yan C, Zhang W. Spatial Distribution and Predictive Significance of Dendritic Cells and Macrophages in Esophageal Cancer Treated With Combined Chemoradiotherapy and PD-1 Blockade. Front Immunol. 2022 Jan 3;12:786429. doi: 10.3389/fimmu.2021.786429. eCollection 2021. PMID 35046943
- [Derived] Zhang W, Yan C, Zhang T, Chen X, Dong J, Zhao J, Han D, Wang J, Zhao G, Cao F, Zhou D, Jiang H, Tang P, Zhao L, Yuan Z, Wang Q, Wang P, Pang Q. Addition of camrelizumab to docetaxel, cisplatin, and radiation therapy in patients with locally advanced esophageal squamous cell carcinoma: a phase 1b study. Oncoimmunology. 2021 Sep 28;10(1):1971418. doi: 10.1080/2162402X.2021.1971418. eCollection 2021. PMID 34616588